CLINICAL TRIAL: NCT02298296
Title: Trajectory of Positive Psychological States in Patients With Acute Coronary Syndrome
Brief Title: Trajectory of Positive Psychological States in Patients With ACS
Acronym: PEACEIIa
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jeff C. Huffman, MD, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2014P000945
Record Dates: First submitted 2014-11-03; First posted 2014-11-21 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment

SUMMARY:
The purpose of the study is to to determine the natural history of positive psychological states, health status, and functioning, over an 8 week period following admission for an acute coronary syndrome (ACS). We aim to compare the changes in these factors from baseline to 8-week follow-up with corresponding changes in the completed proof-of-concept intervention trial (NCT02004158).

ELIGIBILITY:
Inclusion Criteria:

* Suboptimal adherence to health behaviors. This will be defined as mean item score of <15 (suboptimal) on three Medical Outcomes Study-Specific Adherence Scale (MOS SAS) items.
* Submaximal self-reported optimism. This will be defined as a total score of <30 on the Life Orientation Test-Revised (LOT-R) .
* Submaximal self-reported positive affect. This will be defined as a total score of <50 on the Positive and Negative Affect Schedule (PANAS) .

Exclusion Criteria:

* Cognitive deficits, assessed via a 6-item cognitive screen used to assess appropriate participation of medically-ill patients in research studies.
* Medical conditions precluding interviews or likely to lead to death within 6 months, determined in consultation with the primary treatment team and cardiology co-investigator Dr. Januzzi.
* Inability to communicate in English.
* Inability to participate in physical activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects were recruited from inpatient cardiac units in a large, urban hospital.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in positive affect measured by self-report questionnaires | Baseline, 8 weeks
  To determine the change in positive psychological states, specifically optimism and positive affect, over an 8 week period following admission for ACS as measured by the Life Orientation Questionnaire (LOT-R [trait optimism]), Life Orientation Questionnaire-State (LOT-RS [state optimism]), and the Positive and Negative Affect Schedule (PANAS [positive affect]).

SECONDARY OUTCOMES:
Change in behavior adherence measured by a self-report questionnaire | Baseline, 8 weeks
  To assess changes in health behavior adherence over an 8 week period following admission for ACS using the Medical Outcomes Study-Specific Adherence Scale (MOS-SAS items on physical activity, diet, and medication).
Change in function measured by self-report questionnaires | Baseline, 8 weeks
  To assess changes in functional status over an 8 week period following admission for ACS using the Women's Ischemia Syndrome Evaluation (WISE [functional status]) and the Short Form health survey (SF-12 [health-related quality of life]).

CONTACTS AND LOCATIONS:
Overall Officials: Jeff C Huffman, MD, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: No